CLINICAL TRIAL: NCT03501823
Title: Photoacoustic Tomography of Normal and Abnormal Vasculature: Feasibility of in Vivo Measurements.
Brief Title: Development of Photoacoustic Tomography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0248
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Cancer; Cardiovascular Diseases
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peripheral vascular disease: All adult patients (aged 18 years and above) proven or highly suspected to have peripheral arterial or venous disease.
  Ultrasound to be performed first in order to correct Photoacoustic tomography positioning.
  Photoacoustic tomography to be performed after ultrasound
  Interventions: Other: Photoacoustic tomography
- Oncology: All adult patients (ages 18 years and above) proven or highly suspected to have solid organ malignancy Ultrasound to be performed first in order to correct Photoacoustic tomography positioning.
  Photoacoustic tomography to be performed after ultrasound
  Interventions: Other: Photoacoustic tomography

INTERVENTIONS:
Other: Photoacoustic tomography — A non-invasive, safe modality that relies on light and sound to generate images.

SUMMARY:
Cancer is one of the leading causes of death internationally. When planning treatment for most cancers, it is important to know how far it has spread, including whether or not the cancer has spread to the local lymph nodes (LNs) because this affects the treatment strategy. This is termed "staging", and can be achieved by medical imaging, such as by ultrasound, computed tomography (CT) or magnetic resonance imaging (MRI) scans. However, these are imperfect, and sometimes incorrect treatment decisions are made because of errors in staging by imaging. Improved accuracy would be of great clinical value for almost all solid organ tumours. An emerging technique to address this is photoacoustic tomography (PAT), a non-invasive, safe modality that relies on light and sound to generate images. Laser light is applied to the area to be imaged; this is absorbed, and causes the illuminated tissue to emit ultrasound waves. These can be detected and turned into an image by post-processing techniques similar to those used in conventional diagnostic ultrasound. By changing the wavelength of light used, the technique can be adjusted to optimise detection of various body components, including fat, water and both oxygenated and deoxygenated blood. This means the images can represent tissue composition and function rather than just anatomical structure. Hitherto, most work on PAT has been on healthy volunteers, and has focused on imaging the vasculature. We would like to see whether we are able to generate images of deeper structures inside the body. Initially we will focus on patients with vascular disease, whom we expect to have abnormal blood vessels; and subsequently we will attempt to image tumours and LNs in patients with cancer.

DETAILED DESCRIPTION:
Cancer affects nearly 50% of individuals in the UK, and accounts for around 30% of all deaths. For almost all cancers, both prognosis and treatment fundamentally depend on the degree of spread at diagnosis i.e. tumour stage. For example, early stage bowel (colorectal) cancer confined to the bowel wall has a cure rate of nearly 95% whereas it is lower than 50% by the time it has spread to the lymph nodes (LNs). Similarly, patients with LN involvement from breast cancer may require more extensive surgery to remove the affected node, and have poorer long-term survival than patients without LN disease, even with small volumes of nodal tumour. The same is true for most other solid organ malignancies. So, as a general oncological principle, patients with advanced disease often require more aggressive treatment such as pre-operative (neo-adjuvant) chemotherapy, radiotherapy or both; and usually need more extensive surgery / radiotherapy when definitive treatment is instituted.

Such therapeutic decision-making depends fundamentally on the advance knowledge of whether or not a particular patient has disease spread. This, in turn, requires a battery of tests designed to accurately pinpoint the extent and anatomical location of cancer dissemination throughout the body. This is typically achieved via a combination of medical imaging tests (such as ultrasound, computed tomography [CT], magnetic resonance imaging [MRI] and nuclear medicine techniques e.g. positron emission tomography [PET]) and tissue sampling (biopsy). Unfortunately, these techniques are imperfect, both for local staging of the primary cancer and its spread to local LNs. For example, in some cancers, over 50% of malignant LNs measure less than 10mm, the most commonly-used cut-off to define an abnormal lymph node using conventional medical imaging[9]. Therefore, for many tumours it is common practice to treat the entire regional LN group, either by surgical removal or radiotherapy. This strategy risks overtreatment for many and introduces the adverse effects associated with such extensive tissue damage. Regarding primary tumours, the precise extent of local tumour spread can determine whether or not a limited, local resection can be achieved rather than a more radical excision. A rapid, non-invasive, well-tolerated test that could improve local and regional nodal cancer staging would be of great clinical value, since it would immediately permit more accurate individualized treatment strategies.

Photoacoustic tomography (PAT) is a relatively novel technology that may be able to help address this urgent clinical need. PAT relies upon the absorption of laser-generated light of specific wavelengths (often in the infra-red spectrum) by intrinsic components of the imaged tissue. Such absorption results in emission of sound waves, which are ultrasonic (i.e. very high frequency). Images can then be reconstructed in a similar manner to that employed by a clinical ultrasound scanner. By imaging at multiple wavelengths, tissue distribution of water, lipid (fat) and haemoglobin (in red blood cells and therefore blood vessels) can be mapped with extremely high resolution (~100 microns), raising the possibility that PAT can depict the small volume tumour that existing techniques cannot.

ELIGIBILITY:
Peripheral vascular disease:

Inclusion Criteria:

* Adults (aged over 18 years)
* Suspected or proven to have peripheral arterial or venous disease on the basis of physical examination, imaging or ankle-brachial pressure index.
* Able to provide informed consent

Exclusion Criteria:

* Aged 17 or under
* Unable to provide informed consent (e.g. due to dementia or severe mental illness)
* Skin condition precluding safe and/or comfortable placement of an ultrasound or PAT probe (e.g. active infection, ulcerating tumour)

Oncology Cohort All adult patients with either (a) superficial primary tumours or (b) solid organ tumours with a propensity to spread to superficial lymph nodes will be potentially eligible. These include head and neck cancers, breast cancers, skin cancers including melanoma, low rectal and anal cancer, lung cancer and cancers of the upper gastrointestinal tract.

* Adults (aged over 18 years)
* have either a proven diagnosis of malignancy or be under active investigation for malignant disease.
* Able to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially eligible participants will be identified by the direct care clinical team at outpatient clinics, who will inform potential participants of the existence of the study and its broad rationale. Those who wish to consider participation in the study will be provided with a patient information sheet which includes the contact details of the research team.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of PAT acquisitions in which the target lymph node is visible, as judged by the mean of both readers' qualitative scores | 1 year
  Mean score of 2 or above

SECONDARY OUTCOMES:
Dimension of smallest blood vessels resolvable by PAT | 1 year
  Using full-width at half maximum, FWHM, to define the margins of a resolvable vessel

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, London, United Kingdom

REFERENCES:
- [Background] Chen SL, Hoehne FM, Giuliano AE. The prognostic significance of micrometastases in breast cancer: a SEER population-based analysis. Ann Surg Oncol. 2007 Dec;14(12):3378-84. doi: 10.1245/s10434-007-9513-6. Epub 2007 Sep 26. PMID 17899293
- [Background] Zackrisson S, van de Ven SMWY, Gambhir SS. Light in and sound out: emerging translational strategies for photoacoustic imaging. Cancer Res. 2014 Feb 15;74(4):979-1004. doi: 10.1158/0008-5472.CAN-13-2387. Epub 2014 Feb 10. PMID 24514041
- [Background] Guggenheim JA, Allen TJ, Plumb A, Zhang EZ, Rodriguez-Justo M, Punwani S, Beard PC. Photoacoustic imaging of human lymph nodes with endogenous lipid and hemoglobin contrast. J Biomed Opt. 2015 May;20(5):50504. doi: 10.1117/1.JBO.20.5.050504. PMID 26008874
- [Background] Moulding FJ, Roach SC, Carrington BM. Unusual sites of lymph node metastases and pitfalls in their detection. Clin Radiol. 2004 Jul;59(7):558-72. doi: 10.1016/j.crad.2003.12.003. No abstract available. PMID 15208061
- [Background] Zhang E, Laufer J, Beard P. Backward-mode multiwavelength photoacoustic scanner using a planar Fabry-Perot polymer film ultrasound sensor for high-resolution three-dimensional imaging of biological tissues. Appl Opt. 2008 Feb 1;47(4):561-77. doi: 10.1364/ao.47.000561. PMID 18239717